CLINICAL TRIAL: NCT04745741
Title: Evaluating the Rationality of the International Guideline's Recommendations Regarding Selective Coverage of Level Ib in Node Clinical Target Volume With Nasopharyngeal Carcinoma : Results From a Real-world Series
Brief Title: Evaluating the Rationality of the International Guideline About Selective Coverage of Level Ib in CTV With NPC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: NPC006.1
Record Dates: First submitted 2021-02-02; First posted 2021-02-09 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-02

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IB-positive group: Patients with level IB metastasis and histologically confirmed positive by biopsy.
  Interventions: Radiation: IB-positive group

INTERVENTIONS:
Radiation: IB-positive group — The gross tumor volume of the nasopharynx and neck nodes (GTVnx and GTVnd) were delineated according to the tumor extension. The CTVnx was defined as GTVnx + nasopharynx mucosa + 8mm +corresponding anatomical structure without the delineation of CTV1. The CTVnd was defined as GTVnd plus the elective neck area. The prescribe doses of GTVnx/GTVnd, CTVnx, CTVnd were 66-70Gy,54-56Gy and 50-54Gy in 31-35 fractions, respectively.

SUMMARY:
The purpose of this study was to evaluate its rationality in real-world data and provide clinical evidence for the refinement of nodal CTV delineation in nasopharyngeal carcinoma(NPC).

DETAILED DESCRIPTION:
Intensity-modulated radiation therapy (IMRT) has gradually replaced two-dimensional radiation therapy as it offers improved target conformity. Xerostomia is still the most common side effect of radiotherapy in patients with NPC treated with IMRT. Most stimulated saliva is secreted by the parotid glands (PGs), while the submandibular glands (SMGs) produce most of the unstimulated saliva and mucins, which may influence the degree of a dry mouth sensation.There are still differences in the understanding of nasopharyngeal cancer experts at home and abroad on the delineation of clinical target volumes., suitable criteria for elective irradiation of neck level Ib need to be re-evaluated.Therefore, we conducted a retrospective study to assess the feasibility of recommendation to level Ib in the International Guideline for Delineation of Clinical Target Volumes.

ELIGIBILITY:
Inclusion Criteria:

1. histologically confirmed NPC by biopsy (clearly recorded in the pathology report or medical history) ;
2. no evidence of distant metastasis at initial diagnosis and receiving radical IMRT in our center
3. the following conditions: ① level IB metastasis, ② involvement of the submandibular gland, ③ involvement of structures that drain to level Ib as the first echelon site ( the oral cavity, anterior half of nasal cavity involvement) ④ involvement of level II LNs with extracapsular extension（because the judgment of extracapsular invasion is greatly influenced by subjective factors, this study only include patients who had high grade ENE(G2/G3 as demonstrated in our previous study: Oral Oncol. 2019 Dec;99:104438.)⑤ level II nodal involvement with maximum nodal axial diameter greater than 2 cm.
4. all patients who were treated at Lin Shaojun's attending group from June 2005 to December 2012.
5. presence of complete baseline magnetic resonance imaging data of the nasopharyngeal skull base and neck and treated in our center at initial diagnosis .

Exclusion Criteria:

1. disease progression during IMRT;
2. fail to obtain tumor efficacy evaluation information in the medical records of the research center;
3. previous malignancy or other concomitant malignant disease;
4. receiving blind treatment in clinical research.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the inclusion criteria and did not meet the exclusion criteria of our center.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
regional recurrence-free survival (RRFS) | 60 months
  The duration of time to regional failure were calculated from the start of treatment to the dates of recurrence.
level IB nodal recurrence-free survival | 60 months
  The duration of time to level Ib recurrence were calculated from the start of treatment to the date of Ievel Ib recurrence.

SECONDARY OUTCOMES:
local recurrence-free survival (LRFS) | 60 months
  LRFS was calculated from the start of treatment to the dates of local recurrence.
distant metastasis-free survival (DMFS) | 60 months
  DMFS was calculated from the start of treatment to the dates of distant metastasis.
Overall survival | 60 months
  OS was calculated from the date of randomization to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Shaojun Lin, DR, Study Chair — Fujian Cancer Hospital
Locations (1):
- Department of radiation oncology, Fujian cancer hospital, Fuzhou, Fujian, China